CLINICAL TRIAL: NCT04026971
Title: The Effect of Phone Application Supported Nutrition Education on Weight Loss
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ege University (Other)
Responsible Party: Principal Investigator, Doğa Peksever, Registered Dietitian, Ege University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 17-SBE-004
Record Dates: First submitted 2019-04-08; First posted 2019-07-19 (Actual); Last update posted 2019-07-19 (Actual); Status verified 2019-07

CONDITIONS: Obesity
Keywords: obesity; phone application; nutrition education
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Phone Application Supported Nutrition Education (Experimental): Classic nutrition training and diet list is provided. Then notification was sent to obese patients for 3 months by phone application named 'MotiVe'
  Interventions: Procedure: This study is a randomized controlled study aiming to evaluate the effect of phone application supported nutrition education on weight loss according to standard education.
- Classical Nutrition Education (Other): Classic nutrition training and diet list is provided.
  Interventions: Procedure: This study is a randomized controlled study aiming to evaluate the effect of phone application supported nutrition education on weight loss according to standard education.

INTERVENTIONS:
Procedure: This study is a randomized controlled study aiming to evaluate the effect of phone application supported nutrition education on weight loss according to standard education. — This study is a randomized controlled study aiming to evaluate the effect of phone application supported nutrition education on weight loss according to standard education.

SUMMARY:
Internet-based applications are potential supporters for individuals in weight loss programs due to their accessibility and wide access. These applications are aimed at changing the lifestyle of individuals.

This study is a randomized controlled study aiming to evaluate the effect of phone application supported nutrition education on weight loss according to standard education. It has been assumed that the telephone application would increase the adaptation and motivation of the people on diet. Anthropometric measurements and nutritional features of individuals, Weight Efficacy Lifestyle (WEL test), Quality of Life SF-36, Rosenberg Self-Esteem, Obese Individuals Specific Quality of Life, Healthy Life Style Behaviour Scale-II and Healthy Eating Index score changes questioned as intermediate variables. Between March and September 2018, 79 people aged between 18-64 years, whose BMI was 25 and more, who were admitted to the dietitian at Ege University Faculty of Medicine Hospital Endocrine and Metabolic Diseases Clinic and received routine nutrition education were included in the study. In the first interview, the data collection form of all individuals was filled out and anthropometric measurements of all individuals were made by the researcher. All individuals received a classic nutrition education by the clinical dietician and then written personal weight loss diets. Afterwards, only a control appointment for 3 months later was given to the control group. Phone application named Motive designed by the researcher uploaded to only case group's phone. With the telephone application text, visual and video notifications were sent to case group for 3 months.

ELIGIBILITY:
Inclusion Criteria:

* Body mass index is 25 or more.
* Capable of filling the data collection form
* No visual-hearing problems
* Having a smart phone
* Having a internet connection
* Individuals who agreed to participate in the study and whose written consent was obtained

Exclusion Criteria:

* Not having smart phone
* Not having a internet connection
* Those who have undergone bariatric surgery
* Pregnancy
* Thyroid patients that using drugs
* Individuals who require a special diet other than obesity treatment (celiac, gout, diabetes, kidney diseases, coumadin users, etc., diagnosed by a doctor)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 79 (Actual)
Dates: Start 2018-03-01 (Actual); Primary Completion 2018-12-31 (Actual); Study Completion 2018-12-31 (Actual)

PRIMARY OUTCOMES:
Weight Loss | 3 months
  Body weight (kg) was measured at the beginning and end of the study by researcher

SECONDARY OUTCOMES:
Body Mass Index (BMI) | 3 months
  BMI is calculated by dividing the body weight to the height 2 times. Weight was measured with TANITA BC 418 in the clinic. Height was measured with height meter in the clinic. BMI was calculated by researcher at the beginning and end of the study.
Body fat percentage (%) | 3 months
  Body fat percentage was measured with TANITA BC 418, which is available in the clinic by the researcher at the beginning and end of the study .
Waist circumference (cm) | 3 months
  It was measured from the midway of top of hip bone and the bottom of ribs by inelastic tape measure at the beginning and end of the study by researcher.
Neck circumference (cm) | 3 months
  It was measured from just under the larynx at the beginning and end of the study by researcher.
Weight Efficacy Lifestyle (WEL test) | 3 months
  The reliability and validity of the scale has been studied in Turkey. Index was questioned and calculated at the beginning and end of the study by researcher. The increase in the score shows a positive development.
Quality of Life SF-36 | 3 months
  The reliability and validity of the scale has been studied in Turkey. Index was questioned and calculated at the beginning and end of the study by researcher. The increase in the score shows a positive development.
Rosenberg Self-Esteem | 3 months
  The reliability and validity of the scale has been studied in Turkey. Index was questionedand calculated at the beginning and end of the study by researcher. Decreased Rosenberg self-esteem score indicates an increase in self-esteem.
Obese Individuals Specific Quality of Life | 3 months
  The reliability and validity of the scale has been studied in Turkey. Index was questioned and calculated at the beginning and end of the study by researcher. The increase in the score shows a positive development.
Healthy Life Style Behaviour Scale-II | 3 months
  The reliability and validity of the scale has been studied in Turkey. Index was questioned and calculated at the beginning and end of the study by researcher. The increase in the score shows a positive development.
Healthy Eating Index (HEI) | 3 months
  The reliability and validity of the scale has been studied in Turkey. Index was questioned and calculated at the beginning and end of the study by researcher. The increase in the score shows a positive development.

CONTACTS AND LOCATIONS:
Locations (1):
- Ege University, Izmir, TR, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
Internet-based applications are potential supporters for individuals in weight loss programs due to their accessibility and wide access. These applications are aimed at changing the lifestyle of individuals.
  This study is a randomized controlled study aiming to evaluate the effect of phone application supported nutrition education on weight loss according to standard education. It has been assumed that the telephone application would increase the adaptation and motivation of the people on diet. Anthropometric measurements and nutritional features of individuals, Weight Efficacy Lifestyle (WEL test), Quality of Life SF-36, Rosenberg Self-Esteem, Obese Individuals Specific Quality of Life, Healthy Life Style Behaviour Scale-II and Healthy Eating Index score changes questioned as intermediate variables.
Supporting Information: CSR
Time Frame: Access can be opened for an unlimited period of time since the study is published
Access Criteria: Can be examined by researchers working on obesity and applications.